CLINICAL TRIAL: NCT02702219
Title: Effect of Dynamic Flexibility Training Versus Prolonged Static Stretching on Length of the Hamstrings Muscles and Patterns of Lumbar Flexion in Healthy Adults -a Randomized Controlled Trial
Brief Title: Effect of Flexibility Training Versus Static Stretching on Hamstring Muscle Length and Patterns of Lumbar Flexion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luleå Tekniska Universitet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTU_STRETCH_RCT
Record Dates: First submitted 2016-02-26; First posted 2016-03-08 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Static Stretching; Dynamic Stretching; Muscle; Low Back

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dynamic streching (Experimental): Mobility training of the hamstrings muscles to be performed every day
  Interventions: Behavioral: Mobility of the hamstrings muscles
- Static stretching (Active Comparator): Static stretching of the hamstrings muscles to be performed every day
  Interventions: Behavioral: Mobility of the hamstrings muscles

INTERVENTIONS:
Behavioral: Mobility of the hamstrings muscles

SUMMARY:
Mobility training in the form of stretching and flexibility training of our skeletal muscle is a common exercise. However, the evidence are scare and there are only a few studies comparing the effect of prolonged static stretching (> 90 sec) and dynamic flexibility training as to which of these methods has the best length-enhancing effect over time. Further, in clinical practice concerning low back pain, the possibility of a thigh hamstrings muscles to affect movement control of the spine is often mentioned, a link not fully explored in a controlled condition. The purpose of this study is to compare the effect of eight weeks of dynamic flexibility training versus prolonged static stretching on mobility in the hamstring muscles in adults with reduced mobility in the muscles at the back of the thigh. The aim is also to compare the sustained effect of flexibility training between the two groups, eight weeks after completion of the intervention. Furthermore, the aim is to explore how different forms of flexibility training affects movement patterns of the lumbar spine in adult persons with reduced mobility in the hamstrings.

ELIGIBILITY:
Inclusion Criteria:

* Restricted hip flexion < 80 degress due to thight hamstrings muscles

Exclusion Criteria:

* discomfort or illness from musculoskeletal system which significantly affects the person in his/her everyday life
* previous injury (within 12 weeks) in the hamstring muscle prior to study entry
* known RA diagnosis
* known neurological disease
* medication affecting the musculskeletal system

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change of Range of motion of hip flexion | Change from Baseline to after intervention (8 weeks), Change from Baseline to follow-up at 16 weeks
  Hip flexion is performed in a standardised procedure and is measured in degrees.
Change of Fingertip to floor distance | Change from Baseline to after intervention (8 weeks), Change from Baseline to follow-up at 16 weeks
  Distance from fingertip to floor test is performed in a standardised manner and is measured in centimeters

SECONDARY OUTCOMES:
Change in Waiters bow | Change from Baseline to after intervention (8 weeks), Change from Baseline to follow-up at 16 weeks
  Waiters bow is a test of movement controll of the lumbar spine and is measured a if movement is performed correctly or not.
Change in Sitting bilateral knee extension | Change from Baseline to after intervention (8 weeks), Change from Baseline to follow-up at 16 weeks
  Sitting bilateral knee extension is a test of movement controll of the lumbar spine and is measured a if movement is performed correctly or not.

IPD SHARING:
Plan to Share IPD: No